CLINICAL TRIAL: NCT04621968
Title: Correlations Between Nutrition and Urine Spot Checks Via a Urinary Self-test
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Innopsys (Industry)
Collaborators: Centre National de la Recherche Scientifique, France (Other); University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: Innopsys-nurisens-2020
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Diet, Healthy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An inclusion consultation carried out by Professor Gamé at the CHU of Toulouse (Rangueil site) will make it possible to provide the subject with a urinary self-test which automatically carries out and sends the measurement of 10 urinary parameters: pH, density, creatinine, magnesium, calcium, sodium, urea, uric aid, oxalate, citrate.

No samples are taken and therefore stored.

The data will be processed by IRIT in order to investigate :

* the correlation of the analyses with the context of nutrition and sports activity.
* the best recommendation on use (the best time)

Translated with www.DeepL.com/Translator (free version)

DETAILED DESCRIPTION:
Hypothesis We assume that frequent occasional urinary analyses carried out independently by the subject allow us to identify changes in diet.

Final objective:

We would like to determine:

* a strong correlation between the different markers and the nutritional context
* the impact of physical activity on this correlation
* the most relevant moment of analysis (optimising correlation) in order to define recommendations for use

Protocol:

During the inclusion consultation, Professor Gamé will provide the subject's self-test, mobile application and user account. The correspondence table between the user account and the data identifying the subject will only be accessible and kept by Professor Gamé and his team. During this consultation, will be exposed :

* the context and objectives of the study
* the use of the self-test and its recommendations

Thus, no samples will be taken and therefore retained. The cartridges are single-use cartridges and will therefore be thrown away by the subject. The reader will be returned to the partner who developed it (Innopsys) at the end of the protocol.

The subject will have recommendations on the frequency of use which will not be binding and will not have any impact on his participation in the trial. These recommendations will be composed of 2 phases:

Phase 1: frequency of use: 3X/day for 1 month. Phase 2: Frequency of free use. This phase will make it possible to observe the level of acceptability of the technology.

The subject will provide information on his diet by sending a photo of his meals via the mobile application provided. This will then be analysed by algorithms (or operators if the accuracy of the algorithms is insufficient) to extract the type and quantity of food ingested.

Throughout the protocol, the subject will be able to send summary data of his or her sporting activities via the web application linked to the project. These data will be :

* The number of steps taken
* Average heart rate
* The duration of the effort
* The theoretical energy expended

The subject may request a consultation with Professor Gamé during the study in order to have a medical opinion on these results.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

chronic disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers with sport
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
correlation graph between nutrition and urinary measurements | decembre 2020- May 2021